CLINICAL TRIAL: NCT03531060
Title: A Randomised, Double-blind, Placebo-controlled, Phase Ib Study Evaluating the Safety and Tolerability of IRL790 in Patients With Parkinson's Disease (PD) Experiencing Levodopa (L-Dopa) Induced Dyskinesia (LID).
Brief Title: A Clinical Study of IRL790 in Patients With Parkinson's Disease Experiencing Levodopa Induced Dyskinesia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Integrative Research Laboratories AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRL790C002
Record Dates: First submitted 2018-04-10; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — mesdopetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IRL790 (Experimental): IRL790 Capsule 10 mg, oral administration
  Interventions: Drug: IRL790
- Placebo (Placebo Comparator): Placebo capsule, identical appearance, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IRL790 — IRL790 capsule 10 mg
  Arms: IRL790
Drug: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
This is a Phase 1b study investigating the safety and tolerability of IRl790 as adjunct therapy in patients with Parkinson disease. IRL790/placebo is taken for 28 days.

DETAILED DESCRIPTION:
Consenting patients were screened for eligibility as per study-specific inclusion/exclusion criteria within 8-28 days before start of Investigational Medicinal Product (IMP) administration (Visit 1; Screening Visit). At Visit 2 (Day -7) a kinetigraph device (the Parkinson's KinetiGraph™, Global Kinetics Corporation, Melbourne, Victoria, Australia) was attached to the right or left wrist (the parkinsonian dominant side) and baseline patient movement data were recorded during a run-in period of seven consecutive days.

Following baseline assessments at Visit 3 (Day 1) patients were randomized to receive IRL790 or placebo (3:1). The treatment allocation was double-blinded, i.e. it was not disclosed to the patients, the site staff or the Sponsor. During the treatment period, Visits 4-8 were performed on Days 4, 7, 10, 14 and 28 (end of treatment) and a follow-up phone call was performed on Day 21. Dose adjustments of IRL790 could be made until Day 14, following pre-defined criteria. A follow-up visit (Visit 9) was performed 7-10 days after the last IMP dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 50-85 years inclusive.
2. Female patients had to be of non-childbearing potential (defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or post-menopausal females defined as 12 months of amenorrhoea [in questionable cases a blood sample with simultaneous follicle stimulation hormone (FSH) 25-140 IE/L and estradiol <200 pmol/L was confirmatory]).
3. Male patients had to be willing to use condom and contraceptive methods with a failure rate of < 1% to prevent pregnancy7 and drug exposure of a partner and refrain from donating sperm from the date of dosing until three months after dosing of the IMP.
4. A diagnosis of idiopathic PD according to the United Kingdom Parkinson's Disease Society brain bank diagnostic criteria.
5. Showing a clear peak-dose dyskinetic response to regular L-Dopa medication. Patients with additional complex dyskinesia patterns including, but not limited to, diphasic dyskinesias or end of dose dyskinesias could be included if peak dose dyskinesias were also present.
6. On stable doses of anti-parkinson treatment for at least one month prior to inclusion and expected to remain stable on the same doses throughout the study.
7. Clinical laboratory tests within normal limits or clinically acceptable to the Investigator/Sponsor.
8. Able to understand study specific procedures and willing and able to give written informed consent for participation in the study.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, could either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study.
2. History of or present clinically significant psychiatric diagnosis, at discretion of the Investigator.
3. History of seizures, including febrile seizure in childhood.
4. History or presence of hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
5. Any clinically significant illness, medical/surgical procedure or trauma within four weeks of the first administration of IMP.
6. Any planned major surgery within the duration of the study.
7. Previous surgery for PD. . A Hoehn and Yahr score of 5 when "off".

9. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.

10. History of severe allergy/hypersensitivity or on-going allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to IRL790. 11. Administration of another new chemical entity (defined as a compound which has not been approved for marketing) or participation in any other clinical study that included drug treatment with less than three months between administration of last dose and first dose of IMP in this study. 12. History of alcohol abuse and/or use of drugs of abuse. 13. Investigator considered the patient unlikely to comply with study procedures, restrictions and requirements.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 4 weeks
  Medical Dictionary for Regulatory Activities Preferred Term
Physical examination | 4 weeks
  Number of participants with clinically significant abnormal physical examination findings
Electrocardiogram (ECG) recordings | 4 weeks
  Number of participants with clinically significant abnormal electrocardiogram readings
Heart rate | 4 weeks
  Beats per minute
Blood pressure | 4 weeks
  mm Hg
Safety laboratory measurements | 4 weeks
  Number of participants with clinically significant abnormal laboratory values

SECONDARY OUTCOMES:
Unified Dyskinesia Rating Scale (UDysRS) | 4 weeks
  The change from baseline to day 28 of treatment (Visit 4) in the sum of the items comprising the Unified Dyskinesia Rating Scale (UDysRS). The UDysRS is administered to assess dyskinesia. The scoring range is 0-104, where higher score means more dyskinesia.
Unified Parkinson's Disease Rating Scale (UPDRS) | 4 weeks
  The UPDRS assess symptoms of Parkinson's disease. The scoring range from 0-199, where higher score means more severe disease.
Parkinson Kinetigraph (PKG) | Change from run-in to week 4 of treatment
  Wrist worn kinetigraph capturing electronic readings of movement activity.
Clinical Global impression of change (CGI-C) | 4 weeks
  Global impression of change
Pharmacokinetic assessment | 4 weeks
  Plasma concentration at Cmax
Pharmacokinetic assessment | 4 weeks
  Trough level plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Per Svenningsson, MD, PhD, Principal Investigator — Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: No